CLINICAL TRIAL: NCT05879133
Title: HEALTH4CLL2: A Randomized Waitlist Control Trial of Behavioral Interventions in Patients With Chronic Lymphocytic Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: CLL Global Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0411; NCI-2023-04161 (Other: NCI-Clinical Trials Registry)
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Behavioral) (Experimental): Participants are randomly assigned a study group, pariticipants will be given the following:
  * A Fitbit to wear every day during the study. A Fitbit is a physical activity tracking device that will help measure your physical activity. Participants will also receive a Fitbit Aria weight scale. Participants need to create a Fitbit account on the Fitbit website, which will allow participants to track your physical activity and log your diet information and weight. A member of the study team will call you or help you in-person (if you are in the clinic) to help set up the Fitbit and scale.
  * Resistance bands with an instructional video on how to use them.
  * Educational materials, such as handouts about diabetes prevention, as well as written/verbal/video instructions on setting up the Fitbit and scale. This will also include information about online safety/privacy.
  Interventions: Behavioral: Questionnaires; Other: Fit Bit
- Group 2 (Waitlist) (Experimental): Participants are randomly assigned a study group, pariticipants will be given the following:
  * A Fitbit to wear every day during the study. A Fitbit is a physical activity tracking device that will help measure your physical activity. Participants will also receive a Fitbit Aria weight scale. Participants need to create a Fitbit account on the Fitbit website, which will allow participants to track your physical activity and log your diet information and weight. A member of the study team will call you or help you in-person (if you are in the clinic) to help set up the Fitbit and scale.
  * Resistance bands with an instructional video on how to use them.
  * Educational materials, such as handouts about diabetes prevention, as well as written/verbal/video instructions on setting up the Fitbit and scale. This will also include information about online safety/privacy.
  Interventions: Behavioral: Questionnaires; Other: Fit Bit

INTERVENTIONS:
Behavioral: Questionnaires — Survey
Other: Fit Bit — measures physical activity

SUMMARY:
To learn if exercise and weight management can help to improve feelings of fatigue in CLL survivors.

DETAILED DESCRIPTION:
Primary Objective:

--Evaluate the impact of an organized, longitudinal, diet and exercise training program on fatigue as assessed by the Functional Assessment of Cancer Therapy (FACT) score in patients with CLL.

Secondary Objectives:

--Assess changes in physical activity, dietary behavior, physical function using the PROMIS physical function questionnaire and performance tests of physical function, body mass index (BMI) and global quality of life. Additionally, we will assess changes in fecal microbiome composition, metabolic parameters including a comprehensive lipid panel, glucose, insulin, TNF alpha, IL6, leptin, resistin, adiponectin, IGF1 and IGFBP1 and immunologic function as assessed by T cell and monocyte phenotypic and functional assays in patients with CLL after participation in the behavioral intervention.

Exploratory Objectives:

-- Identify differences in the metabolic, immunologic and fecal microbiome composition in patients with CLL who have a high CLL comorbidity index score (CLL-CI) compared to patients with CLL and a low CLL-CI score. And, investigate the association of comorbidity score, disease features, CLL-specific prognostic factors and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-85 years of age with a histologically confirmed diagnosis of CLL and the ability to provide signed informed consent.
* Self-reported physical activity will be assessed prior to enrollment and patients with a physical activity level below the level prescribed in our study will be eligible for inclusion.

Exclusion Criteria:

* Other active malignancy within 1 year of study enrollment (excluding non-melanoma skin cancer)
* Richter's transformation, another medical condition which would prevent safe participation in the behavioral intervention
* Major surgery within 1 month of enrollment
* Non-English speakers
* Cognitively impaired adults
* Pregnancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2027-07-03 (Estimated); Study Completion 2027-07-03 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy (FACT) questionnaires. | through study completion; an average of 1 year.
  Score Scale ranges (0-4)
  0-Not at all
  1-A little bit
  3-Somewhat
  4-Quite a bit
  5-Very much

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferrajoli, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org